CLINICAL TRIAL: NCT06393101
Title: A Randomized, Double-blind, Placebo-controlled Study to Investigate the Effects and Mechanisms of a High CBD Cannabis Extract (BRC-002) for the Treatment of Pain and Health in Complex Regional Pain Syndrome
Brief Title: The Effects and Mechanisms of a High CBD Cannabis Extract (BRC-002) for the Treatment of Pain and Health in Complex Regional Pain Syndrome
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Fadel Zeidan, Associate Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 809767
Record Dates: First submitted 2024-04-24; First posted 2024-05-01 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Complex Regional Pain Syndrome
Keywords: Complex Regional Pain Syndrome; CRPS; Cannabis; Pain
MeSH Terms: conditions — Complex Regional Pain Syndromes; Marijuana Abuse; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo Comparator: 1 Placebo (Placebo Comparator): Half of the patients will receive PO placebo
  Interventions: Drug: BRC-002 Placebo
- Experimental: Active (Experimental): Drug: BRC-002 (High Cannabidiol Botanical Extract) 100 mg/mL
  Interventions: Drug: BRC-002

INTERVENTIONS:
Drug: BRC-002 — BRC-002 is a non-scheduled cannabidiolic (CBD) formulation (<.3% THC). The cannabinoids in BRC-002 are naturally biosynthesized within the Cannabis sativa L. plant as acidic forms of CBD (cannabidiolic acid; CBDA), THC (tetrahydrocannabinolic acid; THCA) and other minor cannabinoids.
  Arms: Experimental: Active
Drug: BRC-002 Placebo — Oral solution of mono-, di-, and triglycerides
  Arms: Placebo Comparator: 1 Placebo

SUMMARY:
The aim of this trial is to determine the potential effects and mechanisms of cannabinoid-induced pain relief in complex regional pain syndrome (CRPS). Multiple psychophysical approaches will be conducted in conjunction with psychological and inflammatory marker testing to determine if and how cannabinoids produce stabilized improvement in CRPS-related pain and comorbidities.

The trial consisted of a pre-treatment screening period, six-week treatment period and a two-week follow-up.

DETAILED DESCRIPTION:
Complex Regional Pain Syndrome (CRPS) is a debilitating and perplexing chronic pain condition that produces incalculable suffering to millions of individuals worldwide. The enigmatic nature of CRPS has left it difficult to treat. CRPS is characterized by a constellation of pain, sensory, autonomic, and motor symptoms that is difficult to pinpoint the source of injury/inflammation. Although unclear, a common cause of CRPS are radial fractures that demonstrate aberrant processing 4-6 weeks after injury.

The aim of this trial is to determine the potential effects and mechanisms of cannabinoid-induced pain relief in complex regional pain syndrome (CRPS). Multiple psychophysical approaches will be conducted in conjunction with psychological and inflammatory marker testing to determine if and how cannabinoids produce stabilized improvement in CRPS-related pain and comorbidities.

The trial consisted of a pre-treatment screening period, six-week treatment period and a two-week follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form.
2. Are between 21-75 years old
3. Ability to communicate in English
4. Volunteers with no previous medical history (e.g., cardiac or pulmonary disease)
5. Are not currently using any type of cannabis, including hemp or CBD
6. Currently 30 days cannabis free
7. Participants with ongoing CRPS [Type 1 or Type 2)] for at least 3 months prior to participation (medical record confirmed)
8. Agrees not to use cannabis, including hemp or CBD, outside of the study during participation in the study
9. Agrees not to use opioids or barbiturates during participation in the study

Exclusion Criteria:

1. Fail cannabis screening
2. Active pulmonary disease
3. Allergy or past adverse effects or negative past experiences from cannabis
4. Positive urine drug test for THC, barbiturates, opioids, oxycodone, or methadone prior to study session 1 or session 2
5. Any significant illness, including cardiovascular disease, diabetes, renal and liver disease
6. Any current or history of an immunocompromising disease or condition (such as lupus, psoriasis, multiple sclerosis, etc.)
7. Any current or history of neurologic conditions, including Parkinson disease, dementia, cognitive impairment, history of seizure disorder, and history of traumatic brain injury/head injury
8. Participant meets DSM-V criteria for current major psychiatric illness, such as bipolar disorder, major depression, psychosis, substance use disorder, or schizophrenia
9. Any current or history of suicidal ideation or attempt
10. Patients with clinically significant laboratory abnormalities

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2029-06-01 (Estimated); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in complex regional pain syndrome pain and heat pain measured with VAS | Day 1 - Day 42
  Change from baseline in pain intensity and unpleasantness ratings using an 11-point Visual Analog Scale in response to heat and ongoing CRPS pain

SECONDARY OUTCOMES:
Pain Inventory Measure | Day 1 - Day 42
  Change from baseline in The Brief Pain Inventory
Depression Measure | Day 1 - Day 42
  Change from baseline in Beck Depression
Sleep Measure | Day 1 - Day 42
  Change from baseline in Pittsburgh Sleep Quality Index
Interleukin 6 | Day 1 - Day 42
  Change from baseline in Interleukin 6

CONTACTS AND LOCATIONS:
Overall Officials: Fadel Zeidan, PhD, Principal Investigator — UC San Diego
Locations (2):
- United States (2):
  - Altman Clinical and Translational Research Institute, La Jolla, California
  - University of California, San Diego, San Diego, California

IPD SHARING:
Plan to Share IPD: No